CLINICAL TRIAL: NCT05366374
Title: Use and Acceptability Study of Swallis DSA™ Device for Distanced Swallowing Assessment for Older Adults In Nursing Home
Brief Title: Use and Acceptability Study of Swallis DSA™ Device for Distanced Swallowing Assessment for Older Adults In Nursing Home CHEZ LES PERSONNES AGEES EN EHPAD
Acronym: SWALL EHPAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Swallis Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-A02894-37
Record Dates: First submitted 2022-04-11; First posted 2022-05-09 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Swallowing assessment with Swallis DSA™ Device — The WALLIS DSA™ investigative device is designed to capture and display pharyngolaryngeal activity in subjects with or at risk of swallowing disorders. The DM is non-invasive: a miniaturized microphone and accelerometer are integrated into the form of a necklace, which will be positioned around the patient's neck to capture the vibroacoustic signals of swallowing during mealtime.

SUMMARY:
SWALL EHPAD is a multicenter, prospective study on the use and Acceptability Study of Swallis DSA™ Medical Device for Distanced Swallowing Assessment for Older Adults In Nursing Home

DETAILED DESCRIPTION:
Swallowing disorders are frequent in nursing homes and under-assessed, under-diagnosed, and under-managed. The SWALLIS DSA™ investigative device is intended to capture and display pharyngolaryngeal activity in subjects with or at risk for swallowing disorders. This device will thus open the way to telecare in the field of swallowing, the expected benefit of which is to improve access to care in the population of subjects living in Nursing Home

This study aims to verify three hypotheses:

1. The recording of the clinical swallowing assessment performed by the speech therapist at a distance allows observation and an interpretation equivalent to the clinical assessment performed in the presence.
2. This device is accepted by all the beneficiaries (residents) and users (nursing staff) in the usual context of a meal situation in a Nursing Home.
3. This device allows the identification of the events marked by the speech therapist and the analysis of the corresponding vibro-acoustic signals.

ELIGIBILITY:
Inclusion Criteria:

* Subject over 60 years old residing in nursing homes
* Subject with a medical prescription for a swallowing assessment
* Subject affiliated or benefiting from the social security system
* Consent to participate obtained in writing and signed by the subject if he/she is able to give his/her consent, or if necessary by the family or, in case of guardianship, by the legally designated representative

Exclusion Criteria:

* Presence of skin lesion(s) on the neck
* Any serious pathology (severe medical condition or behavioral disorder) where, in the opinion of the investigator, it may place participants at additional risk
* Tracheostomized subject
* Subjects with a nasogastric feeding tube
* Subjects under court protection

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: older people living in nursing home diagnosed or suspected of dysphagia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
reproducibility between the swallowing assessment performed in presence and at a distance | up to 6 months
  Comparison of the recommendations resulting from the 2 swallowing assessments carried out by the speech therapist in presence and the speech therapist at a distance on the food adaptations, the assistance with the meals, the need for a check-up or dental care, the adaptation of the environment and the posture

SECONDARY OUTCOMES:
Number of participants who carry the device over the full length of the meal | 1 day
  measurement of the time during which the device is worn
factors that limit the wearing of the device | 1 day
  1. subject's characteristics according to medical history (pathologies, cognitive state, installation and posture)
  2. subjective assessment of difficulty or inability of caregivers to perform the data collection procedure
Quality of the video recording | up to 6 months
  satisfaction scale for the speech therapist

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Ehpad St Jacques, Grenade
  - Ehpad La Résidence, Lisle-sur-Tarn
  - EHPAD L Espérance, Pointis-de-Rivière

IPD SHARING:
Plan to Share IPD: No